CLINICAL TRIAL: NCT04861779
Title: A Phase Ia/b Clinical Study on Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of BTK Protein Degradation Agent HSK29116 in Subjects With Relapsed or Refractory B-Cell Malignancy
Brief Title: A Study of HSK29116 in Adults With Relapsed/Refractory B-cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HSK29116-101
Record Dates: First submitted 2021-04-20; First posted 2021-04-27 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Relapsed/Refractory B-Cell Malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1a Dose Escalation (Experimental): Multiple dose levels of HSK29116 to be evaluated; determination of MTD/Phase 1b recommended dose
  Interventions: Drug: HSK29116
- Phase 1b Dose Expansion in R/R CLL or SLL (Experimental): CLL/SLL patients must have received at least one systemic treatment and failed or relapsed, of which at least half of the subjects must have received covalent BTK inhibitors and have BTK C481 mutation.
  Interventions: Drug: HSK29116
- Phase 1b Dose Expansion in R/R MCL (Experimental): MCL patients must have received at least one systemic treatment and failed or relapsed, of which at least half of the subjects must have received covalent BTK inhibitors and have BTK C481 mutation.
  Interventions: Drug: HSK29116
- Phase 1b Dose Expansion in other R/R B-cell Malignancy (Experimental): Patients must have received at least one systemic treatment and failed or relapsed, of which at least half of the subjects must have received covalent BTK inhibitors and have BTK C481 mutation.
  Interventions: Drug: HSK29116

INTERVENTIONS:
Drug: HSK29116 — Oral HSK29116

SUMMARY:
This is a first-in-human Phase 1a/1b multicenter, open-label oncology study designed to evaluate the safety and anti-cancer activity of HSK29116 in patients with advanced B-cell malignancies.

DETAILED DESCRIPTION:
This study is divided into 2 parts. Phase 1a is a dose escalation to evaluate the safety and tolerability of HSK29116 in adult patients with relapsed/refractory (R/R) B-cell malignancies, who have required and received at least 2 prior systemic therapy and for whom no other therapies are known to provide clinical benefit. Phase 1b will investigate the efficacy of HSK29116 at the dose selected in Phase 1a in up to 3 cohorts of patients with R/R B-cell malignancy indications who have received at least 2 prior systemic therapy：

Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)； Mantle Cell Lymphoma (MCL)； Other B-cell malignancies (they will be selected according to the preliminary results of Phase Ia)

ELIGIBILITY:
Inclusion Criteria:

* Males or females, of any race, aged ≥ 18 years.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0- 2.
* Sufficient bone marrow function, hepatic function and Coagulation function.
* Patients must have measurable disease per disease-specific response criteria.
* Have histologically confirmed R/R CLL,SLL,MCL,Non-GCB DLBCL,FL(grade 1- 3a),MZL,WM.
* Received at least 2 prior systemic therapy and have no other therapies known to provide clinical benefit.
* After the most recent treatment regimen, it is confirmed that PR has not been achieved, or there is confirmed progressive disease.
* Must require systemic therapy.
* The pregnancy test (urine or serum) of female subjects of childbearing potential shall be negative before enrollment.
* Female subjects of childbearing potential and fertile male subjects shall adopt one of the following highly effective contraception measures during the entire study and within 90 days after the study treatment is ended: abstinence, intrauterine device, or hormonal contraceptives beginning at least 3 months before the first dose of IMP.Male subjects are prohibited from donating sperm from the start of study treatment to 90 days after the end of treatment.

Exclusion Criteria:

* Subjects with central nervous system involvement.
* Subjects with histopathological transformation.
* Receipt of allogeneic hematopoietic stem cell transplantation ≤ 180 days before the start of study treatment administration on Cycle 1, Day 1, unless the subject is no longer on immunosuppressant medication. History of autologous hematopoietic stem cell transplantation within 12 weeks (84 days) before the start of study treatment.
* Continuous immunosuppressive therapy, including systemic (such as intravenous or oral) treatment with corticosteroids for the underlying diseases within 2 weeks before the first dose.
* Patients who have received BTKis, tyrosine kinase inhibitors or other targeted small molecule drugs for anti-tumor treatment within 7 days (or 5 half-lives, whichever is shorter) before initiation of study drug; or patients who have received any biological and/or immune-based anti-tumor treatment, including investigational treatment (including but not limited to monoclonal antibody therapy and/or anti-tumor vaccine) within 4 weeks (or 5 half-lives, whichever is shorter); or patients who have received systemic chemotherapy, radiotherapy or traditional Chinese medicines with anti-tumor effect (traditional Chinese medicines with anti-tumor indications specified in the package insert) within 2 weeks (or 5 half-lives, whichever is shorter).
* Previously developed toxicity due to anticancer treatment that did not resolve to Grade ≤ 1 (as per NCI-CTCAE 5.0), except for AEs not constituting a safety risk as assessed by the investigator.
* A history of other malignant tumors within 2 years before enrollment, except for basal cell carcinoma or skin squamous cell carcinoma having been adequately treated, or without disease for ≥ 2 years or with other types of cancer with the survival time of greater than 2 years. Subjects with breast or prostate cancer who are on maintenance hormonal therapies following therapeutic procedures with curative intent are permitted.
* Uncontrolled systemic active infections, or other infections or still on intravenous anti-infection treatment.
* Underwent major surgery in the past 4 weeks.
* Known infection with human immunodeficiency virus, or serologic status reflecting active hepatitis B or C infection.
* Subjects with severe cardiovascular diseases within 6 months before screening.
* Left Ventricular Ejection Fraction < 50% based on either echocardiogram or multigated acquisition (MUGA) scan.
* QTcF ≥ 450 msecs for males and QTcF ≥ 470 msec for females or other significant ECG abnormalities.
* Clinically significant gastrointestinal abnormalities that may affect the intake, transport, or absorption of drugs.
* Requiring or received anticoagulant therapy with warfarin or equivalent vitamin K antagonists (such as phenprocoumon) within 7 days before the first study treatment.
* Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura. Known history of bleeding diathesis.
* A history of stroke or intracranial hemorrhage within 6 months before the first study treatment.
* Use of CYP3A4 inhibitor or inducer within 7 days before the first study treatment, or using of sensitive substrates metabolized by CYP3A4/CYP2B6.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Protocol Specified Dose-Limiting Toxicities | 1 year
  Phase 1a
To establish the MTD and/or recommended Phase 1b dose of HSK29116 | 1 year
  Phase 1a
Number of Participants with Adverse Events and Clinical Laboratory Abnormalities | Up to 3 years
  Phase 1a/1b

SECONDARY OUTCOMES:
Pharmacokinetic(PK) Profile of HSK29116: Maximum Serum Concentration | At the end of Cycle 1 (each cycle is 28 days)
  Phase1a/1b-Sampling of the first dose, pre and post-dose at selected cycle
Overall response rate(ORR) as assessed by the Investigator | Up to 3 Years
  Phase 1a/1b
Duration of response(DoR) as assessed by the Investigator | Up to 3 Years
  Phase 1a/1b
Progression-free survival(PFS) as assessed by the Investigator | Up to 3 Years
  Phase 1a/1b
Time to response(TTR) as assessed by the Investigator | Up to 3 Years
  Phase 1a/1b

CONTACTS AND LOCATIONS:
Overall Officials: Shufang Zhang, Study Director — Haisco Pharmaceutical Group Co., Ltd.
Locations (8):
- One Clinical Research, Perth, Australia
- China (7):
  - NANFANG Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospita, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang